CLINICAL TRIAL: NCT00279864
Title: Prolonged Oral Levofloxacin-Rifampin for Staphylococcus Aureus Prosthetic Joint Infection (PJI) Treated With Debridement And Retention Of Components: A Prospective Observational Cohort Study. Mayo PJI Study Group (MPSG)*
Brief Title: The Utility of Levofloxacin-Rifampin in the Therapy of Prosthetic Joint Infection
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Ortho-McNeil, Inc. (Industry)
Other Study IDs: 415-05; LEVO-BAC-4001
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Staphylococcal Infection; Staphylococcus Aureus Prosthetic Joint Infection
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Prosthetic joint infection is a devastating complication of total joint arthroplasty ultimately leading to the failure of the total joint arthroplasty function and possibly death. Optimal treatment requires the resection of the infected total joint arthroplasty followed by prolonged parenteral antimicrobial therapy. This procedure is followed by reimplantation of a new total joint arthroplasty at a later date. Surgical debridement and retention of the infected total joint arthroplasty offers a more conservative surgical approach and has been proven to be cost-effective in selected groups of patients. Traditional medical therapy for staphylococcal infection would require an initial parenteral antimicrobial followed by chronic oral non-rifampin containing antimicrobial suppression regimen for the life of the total joint arthroplasty. With this strategy the success rate is close to 30%. Recently, several prospective studies of patients with THA, TKA and fracture fixation device infections conducted in Europe showed that the success rate with a 3-6 month course of a quinolone-rifampin combination is effective in 70% to 100% of cases. The proposed study will be a prospective open label observational cohort that will evaluate the outcome of Patients with S. aureus PJI treated with a medical regimen that includes oral levofloxacin- rifampin and debridement and retention of components. This medical regimen was approved for use by the Orthopedic Infectious Diseases focus group, Mayo Clinic, Rochester. 15 patients will be enrolled over a one-year period and followed up to minimum of 1 additional year. The outcome of this group will be compared to a historical group that is treated with traditional therapy.

ELIGIBILITY:
A maximum of 15 adult participants with total hip or total knee arthroplasty are approved for enrollment in this protocol at Mayo Clinic Rochester.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A maximum of 15 adult participants with total hip or total knee arthroplasty are approved for enrollment in this protocol at Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elie F. Berbari, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States